CLINICAL TRIAL: NCT03050385
Title: COgnitive REhabilitation During Transcranial Direct Current Stimulation for Major or Mild Neurocognitive Disorder Patients
Brief Title: Cognitive Rehabilitation During Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2016-048
Record Dates: First submitted 2017-01-03; First posted 2017-02-10 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Transcranial Direct Current Stimulation; Neurocognitive Disorders
Keywords: cognitive rehabilitation
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active stimulation during cognitive rehabilitation (Active Comparator): active transcranial direct current stimulation 20 minutes per session twice a day interval between sessions: more than 20 minutes 7 cm x 5 cm electrodes anodal electrode on F3 cathodal electrode on right forehead 2 mA(milliampere)
  cognitive rehabilitation 10-minute calculation task followed by 10-minute task of local (Japanese) language test
  Interventions: Device: transcranial direct current stimulation
- sham stimulation during cognitive rehabilitation (Sham Comparator): sham transcranial direct current stimulation 20 minutes per session twice a day interval between sessions: more than 20 minutes 7 cm x 5 cm electrodes anodal electrode on F3 cathodal electrode on right forehead 2 mA
  cognitive rehabilitation 10-minute calculation task followed by 10-minute task of local (Japanese) language test
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation

SUMMARY:
The purpose of this study is to explore whether active transcranial direct current stimulation during cognitive rehabilitation tasks can boost cognitive enhancement without severe side effects in mild cognitive impairment or mild dementia patients.

DETAILED DESCRIPTION:
This study explores the additive effect of transcranial direct stimulation compared to sham stimulation during cognitive rehabilitation tasks in mild cognitive impairment or mild dementia patients. Potential participants are recruited by physicians' referral or self-entry. Informed consent by a clinical research coordinator and research physician is performed followed by screening. Participants who passed screening go through 10 sessions of active or sham transcranial direct current stimulation and are evaluated their cognitive function at screening, at the end, and two weeks after the intervention. For quality assurance, independent researcher regularly monitor and audit as participants are enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria:

* participants with a diagnosis of either major neurocognitive disorder or mild neurocognitive disorder, defined in Diagnostic and Statistical Manual of Mental disorder (DSM-5)
* taking the stable dose of psychotropic medication, such as cholinesterase inhibitors or NMDA(N-methyl-D-aspartate) receptor antagonist, for the past two weeks
* ambulant by oneself with or without aiding devices.

Exclusion Criteria:

* with severe psychotic symptoms requiring antipsychotic treatment
* with risks of hospitalization within 6 weeks because of severe depression and/or suicide ideation
* clinically contraindicated to electroconvulsive therapy (ECT) or transcranial direct current stimulation (tDCS)
* with the Mini-Mental State Examination (MMSE) score of less than 18 or the Clinical Dementia Rating Scale (CDR) score of more than 2,
* unable to participate for more than 2 days during the trial
* unable to write a sentence or copy a figure on MMSE at screening.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07-28 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Attrition rate due to adverse events | up to two weeks

SECONDARY OUTCOMES:
difference of Alzheimer Disease Assessment Scale -Cognitive subscale | up to four weeks
  Alzheimer's Disease Assessment Scale - cognitive subscale
difference of the mini mental state examination | up to four weeks
  mini mental state examination
difference of Clinical Dementia Rating scale - sum of boxes | up to four weeks
  Clinical Dementia Rating Scale - sum of boxes
difference of Mini Mental State Examination | up to four weeks
Attrition rate for any reason | up to four weeks
difference of Frontal Assessment Battery | up to four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuma Yokoi, MD, Principal Investigator — NCNP Japan
Locations (1):
- National Center of Neurology and Psychiatry, Kodaira, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inagawa T, Yokoi Y, Narita Z, Maruo K, Okazaki M, Nakagome K. Safety and Feasibility of Transcranial Direct Current Stimulation for Cognitive Rehabilitation in Patients With Mild or Major Neurocognitive Disorders: A Randomized Sham-Controlled Pilot Study. Front Hum Neurosci. 2019 Sep 6;13:273. doi: 10.3389/fnhum.2019.00273. eCollection 2019. PMID 31555109